CLINICAL TRIAL: NCT06269549
Title: Effectiveness of Kinesiological and Dietary Supplement Intervention in Individuals With Knee Osteoarthritis
Brief Title: Kinesiological / Dietary Supplement Intervention in Knee Osteoarthritis
Acronym: KDSKOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Community Healthcare Center dr. Adolf Drolc Maribor (HCM) (Other)
Responsible Party: Principal Investigator, Nejc Sarabon, Full Professor, University of Primorska
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KDS_KOA
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis, Knee
Keywords: exercise; physical activity; dietary supplement
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Intervention Model Description: The differences between groups will be tested using a two-way analysis of variance for repeated measures (factor 1 = group, factor 2 = time)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo blinding / masked for dietary supplement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The effect of dietary supplements added to physical exercise intervention (Other): This study arm will include two groups of participants, one receiving 12 weeks physical exercise intervention together with real dietary supplements (glucosamne and collagen), while the other group receiving exercise intervention with placebo dietary supplements (placebo glucosamine and collagen).
  Interventions: Other: Training Placebo Dietary Supplement (G2); Other: Training Real Dietary Supplement (G3)
- The effect of physical exercise added to dietary supplement intervention (Other): This study arm will include two groups of participants, one receiving 12 weeks real dietary supplements alone (glucosamine and collagen), while the other group receiving real dietary supplements (glucosamine and collagen) with physical exercise.
  Interventions: Other: Non-training Real Dietary Supplement (G1); Other: Training Real Dietary Supplement (G3)

INTERVENTIONS:
Other: Non-training Real Dietary Supplement (G1) — One capsule of glucosamine three times daily, and one packet of hydrolyzed collagen.
  Arms: The effect of physical exercise added to dietary supplement intervention
Other: Training Placebo Dietary Supplement (G2) — One capsule of placebo glucosamine three times daily, and one packet containing placebo collagen + physical exercise (60 minutes per session twice a week)
  Arms: The effect of dietary supplements added to physical exercise intervention
Other: Training Real Dietary Supplement (G3) — One capsule of glucosamine three times daily, and one packet of hydrolyzed collagen + physical exercise (60 minutes per session twice a week)

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of dietary supplement combined with exercise in managing knee osteoarthritis (KOA). The main questions it aims to answer are:

* Is adding a dietary supplement to exercise additionally effective in managing KOA?
* Is adding exercise to the dietary supplement additionally effective in managing KOA?

Participants will be given in three groups:

1. Real dietary supplement alone
2. Real dietary supplement with exercise
3. Placebo dietary supplement with exercise

Investigators will compare groups 1 and 2, or 2 and 3, to answer the research questions.

The hypothesis is that participants who receive the dietary supplement along with exercise will experience greater reduction in pain level, improved physical function, and enhanced quality of life compared to those who receive a placebo combined with exercise or dietary supplement alone.

DETAILED DESCRIPTION:
Participant recruitment will take place at the Community Healthcare Center dr. Adolf Drolc Maribor based on the doctor's recommendation. Following an informed discussion about the study and potential risks, all patients providing written consent will undergo a one-week screening period to determine eligibility for study entry. Upon reaching week 0, patients meeting the eligibility criteria will be randomly assigned in a 1:1:1 ratio to receive either dietary supplements alone, dietary supplements combined with exercise, or placebo dietary supplement combined with exercise.

The effects of the kinesiological / dietary supplement intervention on selected measures will be assessed using a test battery, before and after the 12 week intervention, and at a 6-week follow-up.

Exercise / test batery will be conducted at Community Healthcare Center dr. Adolf Drolc under the supervision of an experienced kinesiologist / investigator.

Based on the posed research questions and hypotheses, investigators would like to highlight the following planned statistical analyses. In the case of bilateral KOA, investigators will analyze the more affected knee for differences between groups. In addition to descriptive statistics, investigators will assess normal distribution and homogeneity of variances. Differences between groups will be tested using two-way repeated measures analysis of variance (factor 1 = group, factor 2 = time) and paired two-tailed post-hoc t-tests with Bonferroni correction. The main comparison will be addressed with a 2x2 two-way analysis of variance. The first research question will be addressed with a 2x2 two-way analysis of variance, including groups 2 and 3. The second research question will be addressed with a two-way analysis of variance, including groups 1 and 2. Additionally, effect size will be calculated. The level of statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis of one or both knee
* severity of knee osteoarthritis based on Kellgren-Lawrence radiographic grade 1-3
* knee pain between 4 and 7 (using a 0-10 scale)

Exclusion Criteria:

* Age <55 years
* Kellgren & Lawrence grade 4 of knee osteoarthritis
* Acute knee injuries within the last 6 months
* Knee pain not associated with knee osteoarthritis
* History of knee or hip endoprosthesis
* Surgery on the back, hip, knee, ankle, or foot within the last 12 months
* Health issues or musculoskeletal limitations affecting strength training and mobility more than knee pain (e.g., lower back pain, hip pain)
* Rheumatoid arthritis, gout
* Neurological conditions (Alzheimer's disease, Parkinson's disease, metabolic diseases affecting the nervous system)
* Muscular or joint diseases/injuries affecting lower limb function (e.g., hip and/or ankle osteoarthritis, sprains, fractures)
* Internal medical conditions (cardiovascular, pulmonary, oncological, diabetes with late complications - diabetic foot, neuropathies) affecting physical performance
* Stroke or similar condition with consequences on motor skills and/or cognition (inability to provide consent)
* Balance disorders, known vestibular system impairment
* Body Mass Index > 32
* Structured strength training exceeding 30 minutes per week
* Corticosteroids and/or hyaluronic acid (intra-articular) use in the last 6 months
* Individuals taking joint health dietary supplements, like glucosamine, chondroitin, or collagen, will need to halt use for at least 30 days before measurements to avoid affecting study outcomes

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in self-assessment pain, stiffness, and physical function (WOMAC questionaire) at week 12 and at a 6-week follow-up | Baseline, week 12 and at a 6-week follow-up
  WOMAC is a self-assessment questionnaire consisting of 24 questions, addressing pain, stiffness, and physical function in individuals with knee or hip osteoarthritis. A higher achieved value or sum of points (0-96) indicates a worse condition.
Change from baseline in self-assessment quality of life (SF-36 questionaire) at week 12 | Baseline and week 12
  SF-36 is a self-assessment questionnaire on quality of life consisting of 36 items, which are grouped into domains measuring eight health components: physical functioning, role limitations due to physical health, role limitations due to emotional health, vitality, mental health, social functioning, bodily pain, and general health. Each item is scored, and each health component provides a score ranging from 0 to 100, where a score of 0 indicates very poor health, while a score of 100 indicates excellent health.
Change from baseline in knee pain on numeric rating scale at week 12 | Baseline and week 12
  Numeric rating scale (NRS) measures pain intensity. It is subjectively assess the current level of knee pain on a scale from 0 (no pain) to 10 (worst possible pain). Change = week 12 score - baseline score
Change from baseline in 40 metre fast-paced walk at week 12 and at a 6-week follow-up | Baseline, week 12 and at a 6-week follow-up
  A timed walk of 4 x 10 metres for a total of 40 metres
Change from baseline in static balance time at week 12 | Baseline and week 12
  A piezoelectric force plate (Kistler, Winterthur, Switzerland, model 9260AA) for a measure forces on the surface, allowing us to record the movement of the center of pressure on the surface over time. The position is a single-leg stance, with the test conducted with eyes open, and parallel stance with the test conducted with eyes open and eyes closed, with three 30-second repetitions in each position. In evaluating the quality of static balance performance, investigators will calculate time of single-leg stance and parallel stance.
Change from baseline in direction-specific amplitude from the center of pressure in static balance at week 12 | Baseline and week 12
  The position is a single-leg stance and parallel stance on piezoelectric force plate (Kistler, Winterthur, Switzerland, model 9260AA) for a measure forces on the surface, with the test conducted with eyes open and eyes closed, with three 30-second repetitions in each position. In evaluating the quality of static balance performance, investigators will calculate overall and direction-specific amplitude from the center of pressure on the surface.
Change from baseline in direction-specific velocity from the center of pressure in static balance at week 12 | Baseline and week 12
  The position is a single-leg stance and parallel stance on piezoelectric force plate (Kistler, Winterthur, Switzerland, model 9260AA) for a measure forces on the surface, with the test conducted with eyes open and eyes closed, with three 30-second repetitions in each position. In evaluating the quality of static balance performance, investigators will calculate overall and direction-specific velocity from the center of pressure on the surface.
Change from baseline in direction-specific frequency from the center of pressure in static balance at week 12 | Baseline and week 12
  The position is a single-leg stance and parallel stance on piezoelectric force plate (Kistler, Winterthur, Switzerland, model 9260AA) for a measure forces on the surface, with the test conducted with eyes open and eyes closed, with three 30-second repetitions in each position. In evaluating the quality of static balance performance, investigators will calculate overall and direction-specific frequency from the center of pressure on the surface.
Change from baseline in number of repetitions in Chair Stand Test at week 12 and at a 6-week follow-up | Baseline, 12 week and at a 6-week follow-up
  Chair Stand Test is measure lower body strength, in which participants stand up repeatedly from a chair for 30 seconds with their arms across their chest. Investigators will measure the number of repetitions in one set.
Change from baseline in time for Five Times Sit to Stand Test at week 12 | Baseline, 12 week and at a 6-week follow-up
  The Five Times Sit to Stand Test scoring is based on the amount of time (to the nearest decimal in seconds) a participant is able to transfer from a seated to a standing position and back to sitting five times with their arms across their chest. Test is used to asses functional lower limbs strength, balance, and fall risk.
Change from baseline in lower body flexibility at week 12 | Baseline and 12 week
  The participant sits on the edge of a chair. One foot must remain flat on the floor, while the other leg is extended forward with the knee straight, heel on the floor, and ankle bent at a 90° angle. One hand is placed on top of the other, with the middle fingers aligned. The participant reaches forward towards the toes by bending at the hips. The back remains straight. The final position is held for 2 seconds. Investigators measure the distance between the fingertips and the toes. Two trials are performed, and the better result is considered.
Change from baseline in Timed up-and-go test (TUG) at week 12 and at a 6-week follow-up | Baseline, week 12 and at 6-week follow-up
  Timed up-and-go test measures functional mobility and balance. Participants will start seated in a chair with armrests. Upon the investigator's signal, participants will rise from the chair, walk 3 meters forward, turn around, walk back to the chair, and sit down. The time taken to complete the task will be recorded to the nearest tenth of a second. The test will be performed three times, and the best time will be recorded for analysis.
Change from baseline in 10-Step Stair Climb Test (SCT) at week 12 and at a 6-week follow-up | Baseline, week 12 and at 6-week follow-up
  After the practice trial, participants will perform one test trial, during which they will be instructed to ascend and descend a flight of 10 stairs as quickly as possible while maintaining safety. The time taken to complete the task will be recorded to the nearest tenth of a second.
Change from baseline in 6-minute walk distance at week 12 | Baseline and 12 week
  6-Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome.
Change from baseline in maximal isometric voluntary contraction of knee flexors and extensors at week 12 | Baseline and week 12
  Maximal isometric voluntary contraction of knee flexion and extension will be performed using a knee dynamometer (S2P, Science in Practice, Ltd., Ljubljana, Slovenia), which will allow knee flexion and extension under static conditions with a knee joint angle of 60° and hip flexion in a seated position at 90°. A support will be placed over the ankle (2-3 cm above the lateral malleolus), through which the participant will press against the measuring part of the device. Before the measurement, the participant will perform two repetitions of flexion and extension with submaximal force, aimed at warming up the participant and familiarizing them with the test requirements. This will be followed by 3 muscle contractions with a 3-second hold at the maximum force produced, during which the participant will be verbally encouraged to achieve maximum strength.

SECONDARY OUTCOMES:
Change from baseline in presence of inflammatory markers in blood sample at week 12 | Baseline and week 12
  Blood sample analysis for the presence of inflammatory markers (CRP, TNF-α, IL-6, IL-1β)
Change from baseline in 24-hour time use at week 12 | Baseline and 12 week
  Assess 24-hour time use with activPAL sensors (sleep, wakefulness, sedentary behavior, physical activity).
Change from baseline in time spent sleeping, awake/sedentary, and physical activity within 24 hour (DAB-Q) at week 12 | Baseline and week 12
  DAB-Q questionnaire for recalling a seven-day period of time use. It assesses the time spent sleeping, awake/sedentary, and engaging in physical activity within the context of 24-hour time use.
Change from baseline in handgrip strength at week 12 | Baseline and week 12
  Handgrip strength will be measured using a hand hydraulic dynamometer. Participants will sit with their elbow flexed at 90° and squeeze the device handle as hard as possible for three seconds. Three repeated measurements will be taken from the dominant hand, and the maximum value (in kilograms) will be recorded.
Change from baseline in number of repetitions in Arm Curl Test at week 12 | Baseline and 12 week
  An arm curl test assess upper body strength. The test involves sitting in a chair holding a weight with the palm facing the body. The arm should be against the trunk to avoid using other muscle groups. As the arm is brought through the range of motion, the wrist should rotate ending up facing the participant (supination). The number of repetitions (as many curls) in 30 seconds is used as the outcome.
Change from baseline in upper body flexibility at week 12 | Baseline and 12 week
  The Back Scratch Test measures how close the hands can be brought together behind the back. This test is done in the standing position. Investigators measure the distance between the tips of the middle fingers. Two trials are performed, and the better result is considered.

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Šarabon, PhD, Study Chair — University of Primorska, Faculty of Health Sciences
Locations (2):
- Slovenia (2):
  - University of Primorska, Faculty of Health Sciences, Izola
  - Community Healthcare Center dr. Adolf Drolc, Maribor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceh T, Zavrsnik J, Sarabon N, Prosen M. Experiences and perceptions of a 12-week combined exercise and dietary supplement program for individuals with knee osteoarthritis: a qualitative focus group study. BMC Musculoskelet Disord. 2026 Jan 20. doi: 10.1186/s12891-026-09509-2. Online ahead of print. PMID 41559644